CLINICAL TRIAL: NCT01007097
Title: A Phase 2, Randomized, Double-Blind, Double-Dummy Placebo-and Active-Controlled, Multicenter Study to Determine the Efficacy and Safety of TAK-875 in Subjects With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of TAK-875 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-875_201; U1111-1111-1019 (Registry Identifier: WHO)
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Non Insulin Dependent; Diabetes Mellitus, Type II; Type 2 Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — TAK-875; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- TAK-875 6.25 mg QD (Experimental)
  Interventions: Drug: TAK-875
- TAK-875 25 mg QD (Experimental)
  Interventions: Drug: TAK-875
- TAK-875 50 mg QD (Experimental)
  Interventions: Drug: TAK-875
- TAK-875 100 mg QD (Experimental)
  Interventions: Drug: TAK-875
- TAK-875 200 mg QD (Experimental)
  Interventions: Drug: TAK-875
- Glimepiride 2 mg or 4mg QD (Active Comparator)
  Interventions: Drug: Glimepiride
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-875 — TAK-875 6.25 mg, tablets and Glimepiride placebo-matching capsules, orally, once daily for up to 12 weeks.
  Arms: TAK-875 6.25 mg QD
Drug: TAK-875 — TAK-875 25 mg, tablets and Glimepiride placebo-matching capsules, orally, once daily for up to 12 weeks.
  Arms: TAK-875 25 mg QD
Drug: TAK-875 — TAK-875 50 mg, tablets and Glimepiride placebo-matching capsules, orally, once daily for up to 12 weeks.
  Arms: TAK-875 50 mg QD
Drug: TAK-875 — TAK-875 100 mg, tablets and Glimepiride placebo-matching capsules, orally, once daily for up to 12 weeks
  Arms: TAK-875 100 mg QD
Drug: TAK-875 — TAK-875 200 mg, tablets and Glimepiride placebo-matching capsules, orally, once daily for up to 12 weeks
  Arms: TAK-875 200 mg QD
Drug: Glimepiride — TAK-875 placebo-matching tablets and Glimepiride 2 mg or 4mg, capsules, orally, once daily for up to 12 weeks.
  Other Names: Amaryl®; Glyree
  Arms: Glimepiride 2 mg or 4mg QD
Drug: Placebo — TAK-875 placebo-matching tablets and Glimepiride placebo-matching capsules, orally, once daily for up to 12 weeks
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine the safety and efficacy of multiple doses of TAK-875, once daily (QD), in subjects with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
TAK-875 is under clinical development for the treatment of type 2 diabetes mellitus in humans. Non-clinical as well as Phase I clinical data suggest that TAK-875 stimulates insulin secretion only at elevated blood glucose levels.

This study is being conducted to study glycemic effects and safety of TAK-875 compared with placebo and glimepiride in subjects with type 2 diabetes who are inadequately controlled on a stable dose of metformin as monotherapy.

Subjects participating in this study are required to fast for 8 hours prior to each study visit, and will be educated in recognition and self-management of hypoglycemia. In addition, during this Run-in Period compliance with study medication will be documented. Subjects who are less than 80% or more than120% compliant with the single-blind, placebo regimen during the run-in period will not be randomized.

At the conclusion of the Run-in period, appropriate subjects will be randomized into the 12 week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Participant meets 1 of the following criteria:

  * A historical diagnosis of type 2 diabetes mellitus without the chronic use of antidiabetic therapy within 8 weeks prior to Screening, and with at least an 8-week documented history of a diet and exercise plan at Screening.
  * A historical diagnosis of mellitus and stable on at least 1500 mg per day or the respective (individually) maximal tolerated dose of metformin as monotherapy for at least 2 months prior to Screening.
* Has a glycosylated hemoglobin level at Screening between 7.5% and 10.0%, inclusive, if on metformin and greater than or equal to 7.5% to less than 11% if treated with diet and exercise alone.
* Has a fasting plasma glucose level less than 260 mg/dL, at Screening.
* Has a fasting C-peptide concentration greater than or equal to 0.8 ng/mL at Screening.
* If participant takes any chronic medications, the dose of these medications must have been stable (no change in dose or drug) for at least 4 weeks prior to Screening.
* Participant's body mass index at Screening is greater than or equal to 23 and less than or equal to 45 kg/m2.
* Is able and willing to monitor glucose with a home glucose monitor and consistently record his or her own blood glucose concentrations.
* Females of childbearing potential who are sexually active must agree to use a medically accepted means of contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study and for 1 month after the last dose of study drug.
* Compliance with single-blind study medication during the Run-in Period is at least 80% and does not exceed 120% based on tablet counts performed by the study staff.

Exclusion Criteria:

* Has systolic blood pressure greater than 160 mm Hg or diastolic pressure greater than 100 mm Hg at Screening or Baseline (as confirmed by repeat measurement 30 minutes after initial measurement).
* Has history of cancer that has been in remission for less than 5 years prior to Screening. A history of basal cell carcinoma or stage 1 squamous cell carcinoma of the skin is allowed.
* Has a creatine phosphokinase level greater than or equal to 5 times the upper limit of normal at Screening.
* Has a hemoglobin level of less than or equal to 12 g/dL (120 gm/L) for men and less than or equal to 10 g/dL (100 gm/L) for women at Screening.
* Has alanine aminotransferase and aspartate aminotransferase levels greater than or equal to 2.5 times upper limit of normal at Screening.
* Has a total bilirubin level greater than or equal to 1.5 mg/dL at Screening.
* The subject has a serum triglyceride concentration greater than or equal to 400 mg/dL at Screening.
* Has an estimated glomerular filtration rate less than or equal to 60 mL/min using the Modification of Diet in Renal Disease equation at Screening.
* Has abnormal thyroid-stimulating hormone levels.
* Has a positive test result for hepatitis B surface antigen or hepatitis C antibody or human immunodeficiency virus.
* Has macro-albuminuria at Screening
* Has a history of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
* Has diabetic gastroparesis that in the investigator's opinion is moderate or severe and hence may impair absorption of study medication.
* Has had coronary angioplasty, coronary stent placement, coronary bypass surgery, myocardial infarction, unstable angina pectoris, clinically significant abnormal electrocardiogram, cerebrovascular accident or transient ischemic attack within 6 months prior or at Screening.
* Has a history of any hemoglobinopathy that may affect determination of glycosylated hemoglobin.
* Received treatment with probucol within 1 year of randomization.
* Donated or received any blood products within 12 weeks prior to Screening.
* Received treatment for more than 7 days within 4 weeks or 8 weeks (depending on the medication) prior to Screening.
* Is on any insulin treatment.
* Received any investigational drug within 4 weeks prior to Screening.
* Is hypersensitive to TAK-875, its excipients or glimepiride.
* Has a history of drug abuse or a history of alcohol abuse within 2 years prior to Screening.
* Has any other physical or psychiatric disease or condition that in the judgment of the investigator may affect life expectancy or may make it difficult to successfully manage and follow the subject according to the protocol.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Probucol
  * Chronically used insulin
  * Chronically used oral or parenteral glucocorticoids
  * Chronically used over-the-counter or prescription weight-loss medications and/or Orlistat Niacin more than 200 mg/day, including niacin-containing products such as Advicor®
  * Chronically used peroxisome proliferator-activated receptor agonists, ezetimibe, oral or injectable hypoglycemic agents other than metformin bile-acid binding agents such as cholestyramine and colesevelam
  * Investigational medications
  * Warfarin and phenytoin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Glycosylated Hemoglobin at Week 12. | Baseline and Week 12

SECONDARY OUTCOMES:
Change from Baseline in Fasting Plasma Glucose at Week 12. | Baseline and Week 12
Change from Baseline in Body Weight at Week 12. | Baseline and Week 12
Incidence of Hypoglycemia During Double-Blind Treatment Period. | Per Occurrence (up to 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (71):
- United States (64):
  - Birmingham, Alabama
  - Hoover, Alabama
  - Tucson, Arizona
  - Anaheim, California
  - Burlingame, California
  - Chula Vista, California
  - Fresno, California
  - Los Angeles, California
  - Los Gatos, California
  - Norwalk, California
  - Orange, California
  - Colorado Springs, Colorado
  - Pueblo, Colorado
  - Boca Raton, Florida
  - Clearwater, Florida
  - Hialeah, Florida
  - Jupiter, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Panama City, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Sandy Springs, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - La Grange, Illinois
  - Sunset, Louisiana
  - Portland, Maine
  - Parkville, Maryland
  - Rockville, Maryland
  - Southfield, Michigan
  - Olive Branch, Mississippi
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Camden, New Jersey
  - West Seneca, New York
  - Asheboro, North Carolina
  - Burlington, North Carolina
  - Charlotte, North Carolina
  - Morehead City, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Carlisle, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Perrysburg, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Altoona, Pennsylvania
  - Tipton, Pennsylvania
  - Cranston, Rhode Island
  - Peak, South Carolina
  - Taylors, South Carolina
  - Varnville, South Carolina
  - Corpus Christi, Texas
  - Hurst, Texas
  - North Richland Hills, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Draper, Utah
  - Salt Lake City, Utah
  - Spokane, Washington
- Guatemala City, Departamento de Guatemala, Guatemala
- Mexico (6):
  - Guadalajara, Jalisco
  - Zapopan, Jalisco
  - Mexico City, Mexico City
  - Cuernavaca, Morelos
  - Monterrey, Nuevo León
  - Tampico, Tamaulipas

REFERENCES:
- [Result] Burant CF, Viswanathan P, Marcinak J, Cao C, Vakilynejad M, Xie B, Leifke E. TAK-875 versus placebo or glimepiride in type 2 diabetes mellitus: a phase 2, randomised, double-blind, placebo-controlled trial. Lancet. 2012 Apr 14;379(9824):1403-11. doi: 10.1016/S0140-6736(11)61879-5. Epub 2012 Feb 27. PMID 22374408